CLINICAL TRIAL: NCT07145606
Title: Effects of Early Rehabilitation Using Blood Flow Restriction and/or Surface Electromyography Biofeedback on Quadriceps Activation and Strength After Anterior Cruciate Ligament Reconstruction: A Multicenter Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole ARC Sante (Other)
Responsible Party: Principal Investigator, Forelli Florian, Assistant Professor ; PhD, Haute Ecole ARC Sante
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMIRACL
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament Injuries; Knee Injuries; Muscle Weakness
Keywords: Anterior Cruciate Ligament; ACL Reconstruction; Knee Injuries; Rehabilitation; Quadriceps Muscle; Quadriceps Activation; Muscle Strength; Arthrogenic Muscle Inhibition; Blood Flow Restriction Training; Surface Electromyography; Biofeedback; Return to Sport
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Muscle Weakness | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Rehabilitation (Active Comparator): Participants receive the standardized postoperative ACL rehabilitation program only. Sessions are supervised approximately 3 times per week for 6 weeks, starting about 2 weeks after surgery. Content includes progressive range of motion, quadriceps activation and strengthening, functional tasks, and return-to-activity progressions delivered per protocol.
  Interventions: Behavioral: Standard Rehabilitation
- Standard Rehabilitation + Blood Flow Restriction (BFR) (Experimental): Participants receive the standardized postoperative ACL rehabilitation plus low-load BFR training. BFR is applied with individualized limb occlusion pressure during prescribed isometric and then dynamic exercises. Sessions are supervised ~3 times per week for 6 weeks beginning ~2 weeks postoperatively.
  Interventions: Behavioral: Blood Flow Restriction (BFR) Training
- Standard Rehabilitation + sEMG Biofeedback (Experimental): Participants receive the standardized postoperative ACL rehabilitation plus surface EMG biofeedback to optimize quadriceps recruitment during targeted tasks (e.g., isometric contractions and functional movements). Real-time visual and/or auditory feedback is provided during supervised sessions ~3 times per week for 6 weeks starting ~2 weeks after surgery.
  Interventions: Behavioral: sEMG Biofeedback
- Standard Rehabilitation + Combined BFR and sEMG Biofeedback (Experimental): Participants receive the standardized postoperative ACL rehabilitation with both adjuncts delivered concurrently: individualized low-load BFR training and sEMG biofeedback during targeted tasks. Sessions are supervised ~3 times per week for 6 weeks beginning ~2 weeks postoperatively.
  Interventions: Behavioral: Blood Flow Restriction (BFR) Training; Behavioral: sEMG Biofeedback

INTERVENTIONS:
Behavioral: Standard Rehabilitation — Standardized postoperative ACL rehabilitation only. Begins ~2 weeks after surgery; supervised ~3 sessions/week for 6 weeks. Includes progressive range of motion, quadriceps activation/strengthening, functional drills, and return-to-activity progressions delivered per protocol.
  Arms: Standard Rehabilitation
Behavioral: Blood Flow Restriction (BFR) Training — Low-load resistance exercises performed with individualized limb occlusion pressure (LOP) determined each session; target %LOP per protocol. Progresses from isometric to dynamic open/closed-chain tasks. Delivered under supervision ~3 sessions/week for 6 weeks; monitoring of tolerance and adverse events per safety LOP.
  Arms: Standard Rehabilitation + Blood Flow Restriction (BFR); Standard Rehabilitation + Combined BFR and sEMG Biofeedback
Behavioral: sEMG Biofeedback — Real-time surface electromyography biofeedback to optimize quadriceps recruitment during targeted tasks (e.g., isometric contractions, straight-leg raise, sit-to-stand, mini-squat, gait drills). Visual and/or auditory feedback with progressive targets. Supervised ~3 sessions/week for 6 weeks; outcome assessors remain blinded.
  Arms: Standard Rehabilitation + Combined BFR and sEMG Biofeedback; Standard Rehabilitation + sEMG Biofeedback

SUMMARY:
Many patients experience quadriceps inhibition after anterior cruciate ligament (ACL) reconstruction, delaying strength recovery, hindering return to sport, and potentially increasing the risk of re-injury. Two rehabilitation strategies-low-load blood flow restriction (BFR) training and surface electromyography (sEMG) biofeedback-aim to enhance neuromuscular activation and strength while limiting joint load. However, comparative and combined evidence in pragmatic, multicenter settings remains limited.

AMIRACL is a multicenter, prospective, randomized, controlled, parallel-group trial with four arms enrolling 200 adults (18-35 years) undergoing a first-time ACL reconstruction. Participants are randomized with center stratification; outcome assessors are blinded to allocation. The four groups are: (1) standard rehabilitation; (2) standard + early BFR; (3) standard + early sEMG biofeedback; and (4) standard + combined BFR and sEMG biofeedback. Interventions begin about 2 weeks postoperatively, are delivered over 6 weeks at three supervised sessions per week, and are integrated into contemporary ACL rehabilitation. BFR uses individualized, auto-regulated cuff pressure during low-load isometric and then dynamic exercises. sEMG biofeedback provides real-time visual and/or auditory feedback to optimize quadriceps recruitment during targeted tasks. The combined arm receives both modalities concurrently.

The primary objective is to compare quadriceps activation (sEMG) and maximal isometric knee extensor strength between groups at 3 and 6 months. Secondary objectives include return-to-sport readiness and patient-reported function (e.g., ACL-RSI, IKDC), broader knee outcomes (e.g., KOOS, Lysholm), adherence and adverse events across arms, and ACL re-injury (ipsilateral graft rupture or contralateral ACL injury) within 2 years. Longer-term patient-reported quality of life is explored up to 5 years.

Key eligibility criteria include age 18-35 years, first ACL reconstruction, and preinjury sport participation; major exclusions include revision ACL surgery, concomitant multi-ligament repair, neuromuscular disorders, and contraindications to BFR or sEMG. The planned sample size is 200 (50 per arm), powered to detect a clinically meaningful between-group difference in quadriceps activation. Analyses will follow the intention-to-treat principle using mixed-effects models for repeated measures. The study is conducted under Good Clinical Practice and applicable Swiss regulations; all participants provide written informed consent. Overall, AMIRACL will determine whether early BFR, sEMG biofeedback, or their combination meaningfully improves quadriceps activation, strength, and clinical recovery after ACL reconstruction compared with standard rehabilitation alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-35 years.

First-time anterior cruciate ligament (ACL) reconstruction.

Pre-injury activity level Tegner ≥ 6.

Marx activity scale ≥ 12.

Body mass index < 35.

With or without associated meniscal injury.

Exclusion Criteria:

* Revision ACL surgery.

Concurrent repair of other knee ligaments.

Neurological or systemic musculoskeletal disorders.

Contraindications to blood flow restriction (BFR) or surface EMG monitoring/biofeedback.

Pregnancy or lactation.

Language barrier or cognitive impairment preventing valid informed consent; vulnerable populations not enrolled.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-04-02 (Estimated); Study Completion 2031-01-02 (Estimated)

PRIMARY OUTCOMES:
Quadriceps neuromuscular activation (surface EMG) | 3 months and 6 months after ACL reconstruction
  Mean normalized surface electromyography (sEMG) activity of the quadriceps during standardized voluntary isometric knee extension; higher values indicate greater activation. Primary analysis compares groups at 3 and 6 months; baseline and post-intervention values are collected to describe trajectories.
Maximal isometric knee extensor strength (traction dynamometry) | 3 months and 6 months after ACL reconstruction
  Peak voluntary isometric knee extension strength recorded with a traction dynamometer under standardized positioning; primary analysis compares groups at 3 and 6 months; baseline and post-intervention values are collected to describe trajectories.

SECONDARY OUTCOMES:
ACL-RSI (Return to Sport after Injury) | 3 months and 6 months after ACL reconstruction
  Patient-reported readiness and psychological response to return to sport using the ACL-RSI questionnaire; higher scores indicate greater readiness.
IKDC (International Knee Documentation Committee) subjective knee form | 3 months and 6 months after ACL reconstruction
  Patient-reported knee symptoms, function, and sports activity; higher scores indicate better status.
ACL re-injury/recurrence rate | 24 months after ACL reconstruction (telephone follow-up)
  Proportion of participants with ipsilateral graft rupture or contralateral ACL injury within 2 years, assessed via structured telephone interview and medical record verification when available.
KOOS (Knee injury and Osteoarthritis Outcome Score) | 5 years after ACL reconstruction
  Patient-reported outcomes across KOOS subscales (Symptoms, Pain, ADL, Sport/Rec, QoL); higher scores indicate better status.
Lysholm Knee Scoring Scale | 5 years after ACL reconstruction
  Patient-reported knee function; higher scores indicate better status.

OTHER OUTCOMES:
Quadriceps neuromuscular activation (sEMG) at end of intervention | Week 8 (post-intervention)
  Normalized sEMG activity measured immediately after the 6-week intervention phase to characterize early neuromuscular changes.
Maximal isometric knee extensor strength at end of intervention | Week 8 (post-intervention)
  Peak isometric knee extension strength measured with traction dynamometry after the 6-week intervention phase to characterize early strength changes.
Adverse events related to rehabilitation and/or BFR/sEMG procedures | Throughout the 6-week intervention and up to Month 6 follow-up
  Number and proportion of participants experiencing adverse events potentially related to the study interventions; categorized by severity (mild/moderate/severe) and seriousness per protocol definitions; events recorded at each supervised session and follow-up visit.

CONTACTS AND LOCATIONS:
Locations (4):
- Orthosport, Domont, France
- Switzerland (3):
  - Movare, Bulle
  - Centre de l'Appareil Locomoteur et du Sport, Hôpitaux Universitaires de Genève (HUG), Geneva
  - Exotherapie, Geneva

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcomes (baseline, Week 8, Month 3, Month 6, and 24-month re-injury status) will be shared, together with a data dictionary and variable codebook. Free-text notes, direct identifiers, and potentially identifying combinations will be removed or masked. Dates will be offset or converted to study days. sEMG raw signals will be shared in anonymized form where feasible.
Supporting Information: Study Protocol, SAP, ICF